CLINICAL TRIAL: NCT07174830
Title: Pharmacokinetic Study of Allisartan Isoproxil Tablets in Healthy Chinese Participants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL065A401
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Allisartan Isoproxil Tablets; safety; tolerability; PK profile
MeSH Terms: interventions — allisartan isoproxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allisartan Isoproxil Tablets 240mg (Active Comparator): Allisartan Isoproxil Tablets 240mg, QD
  Interventions: Drug: Allisartan Isoproxil Tablets 240mg or placebo
- Allisartan Isoproxil Tablets 480mg (Active Comparator): Allisartan Isoproxil Tablets 480mg, QD
  Interventions: Drug: Allisartan Isoproxil Tablets 480mg or placebo
- Allisartan Isoproxil Tablets 720mg (Active Comparator): Allisartan Isoproxil Tablets 720mg, QD
  Interventions: Drug: Allisartan Isoproxil Tablets 720mg or placebo

INTERVENTIONS:
Drug: Allisartan Isoproxil Tablets 240mg or placebo — Allisartan Isoproxil Tablets 240mg or placebo, QD
  Arms: Allisartan Isoproxil Tablets 240mg
Drug: Allisartan Isoproxil Tablets 480mg or placebo — Allisartan Isoproxil Tablets 480mg or placebo, QD
  Arms: Allisartan Isoproxil Tablets 480mg
Drug: Allisartan Isoproxil Tablets 720mg or placebo — Allisartan Isoproxil Tablets 720mg or placebo, QD
  Arms: Allisartan Isoproxil Tablets 720mg

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation study in healthy Chinese subjects at single dose administration of Allisartan Isoproxil Tablets (240 mg ,480 mg or 720 mg）or placebo. The study design allows an assessment of 3 doses with safety monitoring and PK sampling to evaluate the safety, tolerability and PK profile of Allisartan Isoproxil Tablets.

DETAILED DESCRIPTION:
This study will be conducted at 1 study center in Shenzhen. 18 healthy Chinese male and female participants per group, aged 18 to 65 inclusive, will be randomized in a 5:1 ratio to receive a single administration of Allisartan Isoproxil Tablets (240 mg ,480 mg or 720 mg）or placebo (54 participants in total). Each participant will participate in only 1 treatment group. Blood samples will be collected up to 72 hours post-dose for pharmacokinetic parameter calculation, and safety monitoring will continue until sample collection is complete.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults aged 18 to 65 years (inclusive).
* Body weight ≥50 kg for male participants and ≥45 kg for female participants at screening, with a body mass index (BMI) between 19.0 and 25.0 kg/m2.
* Seated systolic blood pressure (SBP) ≥100 mmHg and <140 mmHg, seated diastolic blood pressure (DBP) ≥70 mmHg and <90 mmHg, and no orthostatic hypotension at screening.
* Participants must be able to communicate effectively with the investigator, fully understand the trial's objectives and requirements, voluntarily participate in the clinical trial, and provide written informed consent.

Exclusion Criteria:

* Known or suspected allergy to Allisartan Isoproxil, , other ARBs, or any excipients of this formulation.
* Abnormal findings in physical examination, vital signs, electrocardiogram (ECG), or laboratory tests that are clinically significant as judged by the investigator.
* Any medical history or current condition that may impact participant safety assessments or the pharmacokinetics of the investigational drug, including but not limited to disorders of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, hematologic system, immune system, psychiatric conditions, metabolic abnormalities, or prior gastrointestinal surgery.
* Used any prescription drugs, over-the-counter medications,Chinese herbal medicines, or food supplements within 14 days prior to screening.
* Participants with hyponatremia, hyperkalemia, or hypovolemia;
* Participants with a history of orthostatic hypotension or syncope;
* Participants who have received any vaccinations within 4 weeks prior to screening.
* Participants who consume excessive amounts of strong tea, coffee, and/or caffeinated beverages (≥8 cups/day, 1 cup=250 mL), or have consumed such beverages within 48 hours prior to dosing, or cannot abstain during the trial;
* Participants with habitual intake of xanthine-rich or grapefruit-containing products, or have consumed such products within 48 hours prior to dosing, or cannot abstain during the trial;
* Female participants who are pregnant or breastfeeding;
* Participants (or their partners/spouses) who plan pregnancy, sperm/egg donation, or refuse to use at least one acceptable contraceptive method during the trial and for 3 months post-study ;
* Participants with a positive result for any of the following tests: hepatitis B surface antigen test, hepatitis C antibody test, HIV antibody test, and treponema pallidum antibody test.
* Heavy smokers or Participants with an average tobacco consumption of more than 5 cigarettes per day within 3 months prior to screening, or those who could not completely stop consuming tobacco products during the study.;
* Heavy drinkers or Participants with an average alcohol consumption of more than 14 units per week (1 unit=360 mL beer/45 mL 40% spirits/150 mL wine) within 3 months prior to screening, or with a positive result for breath alcohol test at screening, or those who could not completely stop consuming alcohol-containing food or beverages during the study;
* Participants with a positive result for drug abuse test at screening, or a history of drug abuse(past 5 years), or recent illicit drug use (within 3 months prior to screening);
* Participants who have participated in other drug/device trials and received investigational products within 3 months prior to screening;
* Participants who have donated blood (≥400 mL), received transfusions, or used blood products within 3 months prior to screening;
* Participants with difficult venous access or intolerance to repeated venipuncture;
* Participants with difficulty swallowing study medication; Participants deemed by investigators to have poor compliance or other factors unsuitable for trial participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to Day 4
  Incidence of treatment-emergent adverse events during the whole study
Cmax | Day 1 to Day 4
  Observed maximum plasma concentration (Cmax)
AUC0-t | Day 1 to Day 4
  Plasma concentration-time curve from time zero extrapolated to the time of last quantifiable concentration (AUC0-t)

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Yang, M.D., Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No